CLINICAL TRIAL: NCT00247247
Title: Efficacy and Tolerability of Comtess® Versus Cabaseril® as Add-on to Levodopa in the Treatment of Parkinsonian Patients Suffering From Wearing-Off Phenomenon
Brief Title: Comtess® Versus Cabaseril® as Add-on to Levodopa in the Treatment of Parkinsonian Patients Suffering From Wearing- Off.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2939089; CAMP
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2007-06-25 (Estimated); Status verified 2007-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — entacapone

INTERVENTIONS:
Drug: Comtess®

SUMMARY:
Multi-centre, randomised, parallel-group study, rater-blinded. Total duration of the study per subject is 12 weeks plus a one- to two-week screening period. There are 6 pre-planned visits per subject: screening visit followed by 5 visits. Approximately 300 patients altogether in up to 25 active German study centres and up to 3 active Lithuanian study centres will be randomised.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from idiopathic Parkinson's Disease (PD) with wearing-off phenomenon
* OFF-time per day >= 60 min after the first ON-period in the morning
* 3-5 daily dosages of standard levodopa/DDC inhibitor
* stable antiparkinsonian treatment 3 weeks prior to the randomisation

Exclusion Criteria:

* symptomatic parkinsonism
* concomitant treatment with non-selective MAO inhibitors or a selective MAO-A inhibitor while treated with a MAO-B inhibitor already
* concomitant treatment with one of the following catechol-structured drugs: rimiterol, isoprenaline, adrenaline, noradrenaline, dopamine, dobutamine or apomorphine
* concomitant treatment with alpha-methyldopa, reserpine, typical or atypical neuroleptics, neuroleptic antiemetics (such as metoclopramide) or other drugs with antidopaminergic action
* treatment with COMT-inhibitors 4 weeks prior to the randomisation
* treatment with dopamine agonists 4 weeks prior to the randomisation
* known hypersensitivity to ergot derivatives and entacapone
* dementia (MMSE <= 24)
* depression (Beck Scale >= 17)

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-12; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Primary objective:
- Proof of one-sided equivalence in efficacy regarding the OFF-time (total h of awake time) 12 weeks after start of therapy

SECONDARY OUTCOMES:
Secondary objectives:
- comparison of the tolerability measured as adverse drug reactions in the course of the study
- comparison of the UPDRS total score 12 weeks after start of therapy assessed by a blinded rater
- comparison of the Dyskinesia score 12 weeks after start of therapy assessed by a blinded rater
- comparison of the safety regarding physical examination, vital signs (including blood pressure supine and upright position) and laboratory parameters
- comparison of the results of the disease specific questionnaire PDQ-39
- comparison of clinical global evaluation performed by patient
- comparison of ON-time
- comparison of proportion of ON-time
- comparison of daily levodopa doses and total amount of levodopa
- comparison of daily cabergoline/entacapone doses and total amount of cabergoline/entacapone

CONTACTS AND LOCATIONS:
Overall Officials: Günther Deuschl, Professor, Principal Investigator — Klinikum der Christian-Albrechts-Univeristät zu Kiel
Locations (1):
- Orion Pharma GmbH, Hamburg, Germany